CLINICAL TRIAL: NCT01694368
Title: Multimodality Advanced Intracoronary Imaging With Near-infrared Spectroscopy and Intravascular Ultrasound to Characterize Coronary Artery Plaques Before and After Percutaneous Intervention
Brief Title: Intracoronary Imaging With NIRS-IVUS to Characterize Arterial Plaques
Acronym: NIRS-IVUS
Status: Completed | Type: Observational
Sponsor: Corewell Health West (Other)
Responsible Party: Principal Investigator, Ryan Madder, MD, Physician, Corewell Health West
Other Study IDs: 2011-285
Record Dates: First submitted 2012-09-24; First posted 2012-09-27 (Estimated); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Coronary Artery Disease
Keywords: Near infrared spectroscopy; lipid core; vulnerable plaque
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
To characterize atherosclerotic coronary artery plaques using advanced intra-coronary imaging with a combined near-infrared spectroscopy and intravascular ultrasound catheter before and after percutaneous intervention

DETAILED DESCRIPTION:
This study is being performed to characterize the composition and morphologic characteristics of atherosclerotic coronary artery plaques with intra-coronary near-infrared spectroscopy and intravascular ultrasound in patients undergoing percutaneous coronary intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is at > 18 years of age
2. Subject presents to the catheterization laboratory to undergo clinically-indicated, invasive coronary angiography
3. Subject is willing and able to provide informed written consent
4. Subject is found to have ≥ 1 severe coronary artery stenosis by invasive angiography and percutaneous coronary intervention is planned for definitive treatment or found to have ≥ 1 intermediate coronary artery stenosis and IVUS planned for lesion assessment
5. Coronary anatomy is deemed suitable for combined NIRS-IVUS by the interventional cardiologist performing invasive angiography and intervention

Exclusion Criteria:

1. Subject is pregnant or suspected to be pregnant
2. Subject is unable to provide informed consent
3. Subject has coronary artery anatomy deemed by interventionalist as unsuitable for NIRS-IVUS

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Coronary Artery Disease Patients
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2011-11; Primary Completion 2016-09 (Actual); Study Completion 2021-09 (Actual)

PRIMARY OUTCOMES:
MACCE | 5 year

CONTACTS AND LOCATIONS:
Overall Officials: Ryan D Madder, MD, Principal Investigator — Corewell Health West
Locations (1):
- Spectrum Health; Frederik Meijer Heart &Vascular Institute, Grand Rapids, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Madder RD, Khan M, Husaini M, Chi M, Dionne S, VanOosterhout S, Borgman A, Collins JS, Jacoby M. Combined Near-Infrared Spectroscopy and Intravascular Ultrasound Imaging of Pre-Existing Coronary Artery Stents: Can Near-Infrared Spectroscopy Reliably Detect Neoatherosclerosis? Circ Cardiovasc Imaging. 2016 Jan;9(1):e003576. doi: 10.1161/CIRCIMAGING.115.003576. PMID 26729855